CLINICAL TRIAL: NCT03679689
Title: Improvement of Biochemical Markers After Reduction of Artificially Sweetened Beverages Consumption. A Clinical Randomised Trial
Brief Title: Metabolism Effects of Artificially Sweetened Beverages Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Flores-Muñoz (Other)
Collaborators: Universidad Veracruzana (Other); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor-Investigator, Monica Flores-Muñoz, PhD, Universidad Veracruzana
Organization: Universidad Veracruzana (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D_005/2016
Record Dates: First submitted 2018-09-14; First posted 2018-09-20 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Overweight and Obesity
Keywords: Non-Nutritive sweeteners; Artificially sweeteners; obesity; overweight
MeSH Terms: conditions — Overweight; Obesity | interventions — Artificially Sweetened Beverages

STUDY DESIGN:
Intervention Model Description: A randomized, blind, controlled clinical trial
Who Masked: Investigator
Masking Description: Nobody involved with data acquisition had access to de assignment of the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): no changes in their alimentary habits
- intervention group (Experimental): no intake of artificially sweetened beverages
  Interventions: Dietary Supplement: artificially sweetened beverages

INTERVENTIONS:
Dietary Supplement: artificially sweetened beverages — artificially sweetened beverages restriction
  Arms: intervention group

SUMMARY:
The consumption of artificially sweetened beverages increases glucose and insulin concentrations in blood, body weight and waist circumference. However, the effect of restricting the consumption of these beverages on metabolism is unknown. Our objective is to evaluate the effect of reducing artificially sweetened beverages consumption on the metabolism of overweight and obese young adults. A randomized, blind, controlled 12 week clinical trial will be performed on overweight and obese young adults. Young adults, consumers of artificially sweetened beverages, will be randomly assign to either Control group (no changes in their alimentary habits) or Intervention group (no intake of artificially sweetened beverages). The percentage change between 0 and 12 weeks of anthropometric variables, fasting plasma concentrations of glucose, triglycerides, insulin and cholesterol will be calculated and compared.

DETAILED DESCRIPTION:
Overweight and obesity are public health problems across the world. In 2016 the World Health Organization estimated that over 1900 million adults were diagnosed as overweight or obese. These pathologies result from the interaction between many factors, mainly poor alimentary habits and a sedentary lifestyle. The high consumption of simple carbohydrates and sugar sweetened beverages, like soft drinks, juices and flavored water, is considered one of the main factors that contribute to the increase in incidence and prevalence of overweight and obesity. A high consumption of simple carbohydrates promotes an increase in blood glucose concentrations, which facilitates the formation of triglycerides that are subsequently stored in adipose tissue.

To decrease the caloric intake attributable to sugar sweetened beverages, the food industry promotes the commercialization of artificially sweetened beverages. These products have the same organoleptic features than sugar sweetened beverages, with the perks of having a minimum or no caloric contribution at all, not affecting the energy metabolism.

Nonetheless, recent studies relate the consumption of artificially sweetened beverages with a deregulation of the metabolic homeostasis, promoting physiological modifications. Likewise, it was reported that artificial sweeteners increased glucose and insulin concentrations in blood, which is detrimental to health, especially in population with a pre-existing risk of developing non-infectious diseases, such as overweight and obesity. For this reason we will evaluate the effect of reducing the consumption of artificially sweetened beverages (ASBs) in overweight and obese young adults.

This study is a single-blind randomized clinical trial controlled with a parallel group. Young adults, students of the University of Veracruz, are randomly allocated to a 12-week no consumption of artificially sweetened beverages intervention or control group.

All the volunteers that satisfy the inclusion criteria will be asked to sign the informed consent before the start of the study. The volunteers will be randomly allocated in control or intervention group (1:1 allocation ratio to each group) in blocks of 2 using Microsoft Office Excell. Nobody involved with data acquisition will have access to the assignment of the participants. Once randomly assigned, a blood sample and anthropometric variables will be taken to establish basal data. Participants will be interviewed to know caloric intake (24-h food recall), consumed portions and beverage consumption (Food frequency questionnaire). The intervention group will not be allowed to consume artificially sweetened beverages; however, they will be allowed to consume products that do not contain artificial sweeteners in their formulae. For the control group artificially sweetened beverages consumption will not be modified. Both groups will continue with their normal food habits. Anthropometric measures, 24-h food recall and food frequency questionnaire data will be collected at week 0, 6 and 12. A blood sample will be taken at week 0 and 12. In order to categorize the physical activity a, previously validated, questionnaire will applied. Using this instrument, physical level will be divided in low, moderate and high.

For comparison between groups at baseline measurements we will use Student´s t-test and Mann- Whitney U test based on data distribution. In order to compare changes between baseline and 12 weeks measurements, the percentage change will be calculate, and pertinent tests applied. A p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 kg /m² to 36 kg / m², with low intensity physical activities and consumers of at least 3 portions of artificially sweetened beverages per week

Exclusion Criteria:

* students with hyper or hypothyroidism, pregnant women and those who perform high to moderate physical activities

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Glucose in mg/dl | 12 weeks
  Fasting blood samples will be analyzed for plasma concentrations
Triglycerides in mg/dl | 12 weeks
  Fasting blood samples will be analyzed for plasma concentrations
Insulin | 12 weeks
  Fasting blood samples will be analyzed for plasma concentrations
Cholesterol in mg/dl | 12 weeks
  Fasting blood samples will be analyzed for plasma concentrations

SECONDARY OUTCOMES:
Micro and macronutrients consumed during the 12 week study (in grams) | 12 weeks
  24-hour recall
Weight in kilograms | 12 weeks
  bioelectrical impedance
Body fat percentage | 12 weeks
  bioelectrical impedance
Portions consumed of artificially sweetened beverages (1portion=250ml) | 12 weeks
  food frequency instrument

CONTACTS AND LOCATIONS:
Overall Officials: Monica Flores-Muñoz, PhD, Study Director — Universidad Veracruzana
Locations (1):
- Universidad Veracruzana, Xalapa, Veracruz, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergwall S, Johansson A, Sonestedt E, Acosta S. High versus low-added sugar consumption for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2022 Jan 5;1(1):CD013320. doi: 10.1002/14651858.CD013320.pub2. PMID 34986271

DOCUMENTS (1):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03679689/Prot_000.pdf